CLINICAL TRIAL: NCT00928629
Title: Audit and Screening Study to Determine the Prevalence of Peripheral Arterial Disease. A Cross-sectional Multi-centre Clinical Study in Subjects With Cardiovascular Disease Risk Factors.
Brief Title: Audit and Screening Study to Determine the Prevalence of Peripheral Arterial Disease
Acronym: ACHILLES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Pretium Pty Ltd (Unknown)
Responsible Party: MC MD, AstraZeneca
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: D3560L00089
Record Dates: First submitted 2009-06-23; First posted 2009-06-26 (Estimated); Last update posted 2009-11-13 (Estimated); Status verified 2009-11

CONDITIONS: Peripheral Arterial Disease
Keywords: Peripheral Arterial Disease; Cardiovascular Disease; Vascular Disease
MeSH Terms: conditions — Peripheral Arterial Disease; Cardiovascular Diseases; Vascular Diseases | interventions — Mass Screening

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All Subjects (Other): ABI Screening Test Population: Subjects of either sex, any race, with at least two of the specified CVD risk factors, with no overt cardiovascular disease.
  Interventions: Procedure: Ankle-brachial index (ABI) Screening Test

INTERVENTIONS:
Procedure: Ankle-brachial index (ABI) Screening Test — Patients will undergo an ABI measurement

SUMMARY:
The primary objective of the study is to establish the prevalence of lower extremity peripheral arterial disease (PAD), defined as an ankle-brachial index of less than or equal to 0.9, in subjects with at least two of the specified cardiovascular disease (CVD) risk factors, with no overt cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

* Males aged 45 years or above or females aged 55 years or above (age related CVD risk factor).
* At least two other risk factors for CVD: cigarette smoking, diabetes mellitus, hypertension, low HDL or high LDL cholesterol, strong family history of coronary heart disease, elevated waist circumference, Aboriginal and/or Torres Strait Islander.
* Willingness to participate in study and sufficient command of the English language to read and complete study questionnaire.

Exclusion Criteria:

* Less than 2 risk factors for CVD (other than age), symptoms of PAD, coronary heart disease or coronary heart disease risk equivalents
* No lipid data collected in the last 12 months
* Serious or unstable medical or psychological conditions that, in the opinion of the Investigator, would compromise safety or successful participation in the study.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2009-06; Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Prevalence of lower extremity peripheral arterial disease, defined as an ankle-brachial index of < or = 0.9 in subjects with at least two of the specified CVD risk factors, with no overt cardiovascular disease | 1 visit

SECONDARY OUTCOMES:
Prevalence of cardiovascular risk factors in the target population | 1 visit
Cardiovascular risk level and cardiovascular risk factor management in the target population pre and post study | 1 visit
Subject characteristics that are determinants of PAD diagnosis | 1 visit

CONTACTS AND LOCATIONS:
Overall Officials: Simon Fisher, Study Director — AstraZeneca; Amelia Siu, Study Director — AstraZeneca; David Sullivan, Principal Investigator — Central Clinical School, The University of Sydney, Sydney, Australia
Locations (23):
- Australia (23):
  - Research Site, Edgecliff, New South Wales
  - Research Site, Hinchinbrook, New South Wales
  - Research Site, Kingsford, New South Wales
  - Research Site, Kingswood, New South Wales
  - Research Site, Liverpool, New South Wales
  - Research Site, Mosman, New South Wales
  - Research Site, Neutral Bay, New South Wales
  - Research Site, Sydney, New South Wales
  - Research Site, Aspley, Queensland
  - Research Site, Morayfield, Queensland
  - Research Site, Parkwood, Queensland
  - Research Site, Beulah Park, South Australia
  - Research Site, Glenelg East, South Australia
  - Research Site, Surrey Downs, South Australia
  - Research Site, Bridgewater, Tasmania
  - Research Site, Kingston, Tasmania
  - Research Site, Sandy Bay, Tasmania
  - Research Site, Brighton, Victoria
  - Research Site, Lalor, Victoria
  - Research Site, Preston, Victoria
  - Research Site, Booragoon, Western Australia
  - Research Site, East Victoria Park, Western Australia
  - Research Site, Woodvale, Western Australia